CLINICAL TRIAL: NCT05926687
Title: Optimizing Outcomes Through Sequencing Parent-Mediated Interventions for Young Children With Autism
Brief Title: Optimizing Outcomes for Young Autistic Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Megan Roberts, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: STU00216950
Record Dates: First submitted 2023-06-07; First posted 2023-07-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: intervention; early intervention; toddlers; autistic; autism; virtual; tele-health
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The investigators propose a sequential, multiple assignment, randomized trial (SMART) design in which the investigators will initially randomly assign 184 children with ASD, between 18 and 48 months of age, to receive either the SC or DB intervention. Following each respective manualized, 12-week intervention (first-stage intervention; SC or DB), the interventionist will measure the parents' use of intervention strategies. At this point, all parents will be re-randomized before starting the second-stage intervention. Participants will be re-randomized to receive the same intervention at a lower frequency (Reduce) or to receive the other intervention (Switch). Parents who need additional parent instructional method, such as video feedback will be randomized to receive additional tools (Augment).
Who Masked: Outcomes Assessor
Masking Description: Outcome coders will be blind to experimental condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Social Communication + Reduce Frequency (Active Comparator): Starting Intervention: Social Communication Who: Parent & Child & Therapist Frequency: 1-hour twice/week
  Secondary Intervention: "Reduce Frequency" of Social Communication Intervention Intervention: Social Communication Who: Parent & Child & Therapist Reduce Frequency: 1-hour once/week
  Interventions: Behavioral: Social Communication; Behavioral: Social Communication + Reduce Frequency
- Social Communication + Add Tools (Active Comparator): Starting Intervention: Social Communication Who: Parent & Child & Therapist Frequency: 1-hour twice/week
  Secondary Intervention: "Add Tools" to Social Communication Intervention Intervention: Social Communication Who: Parent & Child & Therapist Frequency: 1-hour twice/week Add: Video feedback
  Interventions: Behavioral: Social Communication; Behavioral: Social Communication + Add Tools
- Social Communication + Switch Intervention to Disruptive Behavior (Active Comparator): Starting Intervention: Social Communication Who: Parent & Child & Therapist Frequency: 1-hour twice/week
  Secondary Intervention: Switch to Disruptive Behavior Intervention Who: Parent & Therapist only Frequency: 1-hour once/week
  Interventions: Behavioral: Social Communication; Behavioral: Disruptive Behavior
- Disruptive Behavior + Reduce Frequency (Active Comparator): Starting Intervention: Disruptive Behavior Who: Parent & Therapist only Frequency: 1-hour once/week
  Secondary Intervention: "Reduce Frequency" of Disruptive Behavior Intervention Intervention: Disruptive Behavior Who: Parent & Therapist only Reduce Frequency: 1-hour every other week
  Interventions: Behavioral: Disruptive Behavior; Behavioral: Disruptive Behavior + Reduce Frequency
- Disruptive Behavior + Add Tools (Active Comparator): Starting Intervention: Disruptive Behavior Who: Parent & Therapist only Frequency: 1-hour once/week
  Secondary Intervention: "Add Tools" to Disruptive Behavior Intervention Intervention: Disruptive Behavior Who: Parent & Therapist & Child Frequency: 1-hour once/week Add: Video feedback
  Interventions: Behavioral: Disruptive Behavior; Behavioral: Disruptive Behavior + Add Tools
- Disruptive Behavior + Switch Intervention to Social Communication (Active Comparator): Starting Intervention: Disruptive Behavior Who: Parent & Therapist only Frequency: 1-hour once/week
  Secondary Intervention: "Switch" to Social Communication Intervention Who: Parent & Child & Therapist Frequency: 1-hour twice/week
  Interventions: Behavioral: Social Communication; Behavioral: Disruptive Behavior

INTERVENTIONS:
Behavioral: Social Communication — Intervention: Social Communication Who: Parent & Child & Therapist Frequency: 1-hour twice/week
  Other Names: SC; Project Impact
  Arms: Disruptive Behavior + Switch Intervention to Social Communication; Social Communication + Add Tools; Social Communication + Reduce Frequency; Social Communication + Switch Intervention to Disruptive Behavior
Behavioral: Disruptive Behavior — Intervention: Disruptive Behavior Who: Parent & Therapist only Frequency: 1-hour once/week
  Other Names: RUBI; DB
  Arms: Disruptive Behavior + Add Tools; Disruptive Behavior + Reduce Frequency; Disruptive Behavior + Switch Intervention to Social Communication; Social Communication + Switch Intervention to Disruptive Behavior
Behavioral: Social Communication + Reduce Frequency — Intervention: Social Communication Who: Parent & Child & Therapist Frequency: 1-hour once/week
  Arms: Social Communication + Reduce Frequency
Behavioral: Social Communication + Add Tools — Intervention: Social Communication Who: Parent & Child & Therapist Frequency: 1-hour twice/week
  Arms: Social Communication + Add Tools
Behavioral: Disruptive Behavior + Reduce Frequency — Intervention: Disruptive Behavior Who: Parent & Therapist only Frequency: 1-hour every other week
  Arms: Disruptive Behavior + Reduce Frequency
Behavioral: Disruptive Behavior + Add Tools — Intervention: Disruptive Behavior Who: Parent & Therapist only Frequency: 1-hour once/week
  Arms: Disruptive Behavior + Add Tools

SUMMARY:
The overarching goal of the proposed study is to: (a) determine how best to sequence two parent-mediated interventions: a social communication intervention (Project ImPACT, Improving Parents as Communication Teachers) and a disruptive behavior intervention (Parent Training for Disruptive Behavior) and (b) examine moderators and mediators of intervention outcomes.

DETAILED DESCRIPTION:
Despite advances in early identification of and intervention for children with autism spectrum disorders (ASD), the long-term outcomes for children with ASD remain variable. As many as 40% of children with ASD are minimally verbal at 9 years of age, and 75% of adults with ASD have persistent social communication (SC) difficulties. Furthermore, as many as 70% of children with ASD have a co-occurring diagnosis of disruptive behavior (DB) disorder. Parents play an important role in SC development and in the prevention of and intervention for DB. As such, the overarching goal of the proposed study is to: (a) determine how best to sequence two parent-mediated interventions: an SC intervention (Project ImPACT, Improving Parents as Communication Teachers) and a DB intervention (Parent Training for Disruptive Behavior) and (b) examine moderators and mediators of intervention outcomes. While evidence of efficacy and feasibility exist for both of these interventions individually, an adaptive intervention approach that considers and optimizes both interventions has not been evaluated. This type of adaptive intervention approach may be particularly needed in parent-mediated interventions due to the cost, burden, and complexity of teaching parents to use multiple intervention strategies. To determine the optimal intervention sequence that considers parent moderators and parent use of intervention strategies, the investigators propose a sequential, multiple assignment, randomized trial (SMART) design in which the investigators will initially randomly assign 184 children with ASD, between 18 and 48 months of age, to receive either the SC or DB intervention. Following each respective manualized, 12-week intervention (first-stage intervention; SC or DB), the interventionist will measure the parents' use of intervention strategies. At this point, all parents will be re-randomized before starting the second-stage intervention. Second-stage intervention decisions are designed to be responsive to parents' implementation of the first-stage intervention strategies. That is, parents who are implementing the first-stage intervention strategies with high fidelity (high implementers) will be re-randomized to receive the same intervention at a lower frequency (Reduce) or to receive the other intervention (Switch). Parents who are implementing the first-stage intervention strategies with low fidelity (low implementers) will be re-randomized to receive the same intervention with an additional parent instructional method, such as video feedback (Augment) or to receive the other intervention (Switch). After 24 weeks of intervention (12 weeks for first stage, 12 weeks for second stage), the investigators will assess child SC skills, child DB, and family life participation in everyday activities. The investigators will also measure parent-child joint engagement continually during intervention to examine the extent to which joint engagement mediates intervention outcomes. The proposed research is significant because if an intervention for one domain (SC or DB) has an impact on the other, an intervention sequence that systematically includes both interventions may have an even greater impact on both domains.

ELIGIBILITY:
Inclusion Criteria:

* Child is between 18 and 48 months old
* Child scores above the research cutoff for ASD on the TELE-ASD-PEDS
* Child has no other known diagnosis or disability at study entry
* Child has normal vision
* Child is exposed to English at least 50% of the time
* Child has a caregiver willing to learn the intervention strategies
* Caregiver wants help supporting their child's social communication and behavior regulation
* Caregiver understands conversational English well enough to participate in caregiver instruction

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 184 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Observed Child Social Communication | Between 25-30 weeks
  The child's observed social communication is measured from a caregiver-child interaction in which the dyad interacts across a variety of daily activities using materials in their home. This interaction will be recorded and coded for the child's social communication using the codebook from the Early Communication Indicator assessment.
Observed Child Disruptive Behavior | Between 25-30 weeks
  The child's disruptive behavior is measured from a caregiver-child interaction in which the dyad interacts across a variety of daily activities using materials in their home. This interaction will be recorded and coded for the child's disruptive behavior using the Disruptive Behavior Diagnostic Observation (DB-DOS) codebook.
Caregiver Report of Child Social Communication | Between 25-30 weeks
  The caregiver's assessment of the child's social communication is measured from the Developmental Profile 4 (DP-4) Social-Emotional and Communication Scales. This assessment will yield a total raw score ranging from 0 (minimum) to 70 (maximum), with higher scores indicating better outcomes.
Caregiver Report of Child Disruptive Behavior | Between 25-30 weeks
  The caregiver's assessment of the child's disruptive behavior is measured from the Eyberg Child Behavior Inventory.
Family Life Impairment Scale | Between 25-30 weeks
  Family life participation outcomes are measured using the Family Life Impairment Scale. The measure's values range from 0 (minimum) to 38 (maximum) with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
Caregiver Satisfaction | Between 25-30 weeks
  The caregiver's satisfaction with the intervention(s) are measured from a researcher developed satisfaction questionnaire. Sample items include asking about the caregiver's confidence in supporting their child's development, the difficulty in finding time to support their child's development, the added stress of participating in the study, the reasonableness of the study time requirement, the satisfaction with their study therapist's presentation of the material, and whether they would recommend the intervention to another family.
Caregiver Perceived Stress | Between 25-30 weeks
  The caregiver's stress levels are measured using the Perceived Stress Scale. The measure's values range from 0 (minimum) to 40 (maximum) with higher scores indicating worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the final dataset in two ways: the National Database for Autism Research (NDAR) and the Inter-University Consortium for Political and Social Research (ICPSR).
Supporting Information: Study Protocol
Time Frame: Data will be shared once the first published article is available. Data will be available for 10 years.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT05926687/Prot_ICF_000.pdf